CLINICAL TRIAL: NCT03453177
Title: Intravenous and Oral Fosfomycin in Hospitalised Neonates With Clinical Sepsis: an Open-label Safety and Pharmacokinetics Study (neoFosfo)
Brief Title: Intravenous and Oral Fosfomycin in Hospitalised Neonates With Clinical Sepsis
Acronym: NeoFosfo
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Drugs for Neglected Diseases (Other)
Collaborators: KEMRI-Wellcome Trust Collaborative Research Program (Other); University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Neo-Fos-001
Record Dates: First submitted 2018-02-07; First posted 2018-03-05 (Actual); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Neonatal SEPSIS
MeSH Terms: conditions — Neonatal Sepsis | interventions — Standard of Care; Fosfomycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard of Care (No Intervention): ampicillin 50mg/kg twice daily and gentamicin [3mg/kg for babies <2kg or 5mg/kg for babies >2kg] once daily for 7 days, as per Kenyan guidelines).
- Standard of Care plus Fosfomycin (Experimental): Fosfomycin will initially be administered IV for at least 48 hours together with standard care (ampicillin + gentamicin). Then, once babies are tolerating oral feeds and clinically improved, fosfomycin will be changed to oral administration to complete a total of 7 days of fosfomycin (or until the baby is discharged).
  Interventions: Drug: Standard of Care + Fosfomycin; Procedure: PK; Procedure: Analysis of Bacterial Isolates

INTERVENTIONS:
Drug: Standard of Care + Fosfomycin — Fosfomycin will initially be administered IV for at least 48 hours together with standard care (ampicillin + gentamicin). Then, once babies are tolerating oral feeds and clinically improved, fosfomycin will be changed to oral administration to complete a total of 7 days of fosfomycin (or until the baby is discharged).
  Other Names: iv Fosfomycin; oral Fosfomycin
  Arms: Standard of Care plus Fosfomycin
Procedure: PK — Two PK samples will be taken after each of the first IV and oral doses, with sampling times allocated within possible early (5, 10 or 60 minutes) and late (2, 4 or 8 hours) time-points after starting the IV and PO formulations; then again together with biochemistry after 7 days for those babies whom remain as inpatients.
  Arms: Standard of Care plus Fosfomycin
Procedure: Analysis of Bacterial Isolates — For assessment of susceptibility patterns in bowel flora, we will systematically assess all admission and discharge nappy swabs.
  Arms: Standard of Care plus Fosfomycin

SUMMARY:
Neonatal sepsis has a high risk of morbidity and mortality. The current WHO and national guidelines recommend antibiotics to which resistance is reported in neonatal populations, although the available data is limited. Research on alternative empirical regimens for neonatal sepsis which are affordable, safe and cost-effective, with a step-down oral option, is needed. AMR is an issue of global public health concern and is one of the WHO's global health priority areas. Understanding the benefits, risks, MIC capacity and PK of fosfomycin will influence global policy on the case management of neonates with sepsis in Kenya and international settings.

DETAILED DESCRIPTION:
Antimicrobial resistance (AMR) has become a major issue in global health. Despite progress in the reduction of under 5 mortality rates in recent decades, the proportion of neonatal deaths occurring within this age group has increased, with almost one quarter of all neonatal deaths occurring due to serious bacterial infection. Common bacteria causing neonatal sepsis are now exhibiting widespread resistance to several classes of antibiotics. There is an urgent need to discover new, effective treatments and re-evaluate existing therapeutic agents to treat infections potentially caused by multi-drug resistant (MDR) pathogens. Gram-negative bacteria (GNB) predominate as the cause of neonatal sepsis, and are increasingly associated with high rates of resistance to the currently recommended WHO empirical therapy regimen of ampicillin/penicillin and gentamicin. There is therefore a need to develop an updated empiric regimen with improved efficacy in the context of increasing MDR sepsis in neonates. New antimicrobials under development will be expensive once licensed, and there are currently virtually no planned trials to assess their efficacy in neonates in low- and middle-income countries (LMICs).

One potential strategy is utilising an existing off-patent (and therefore affordable) antibiotic available in intravenous and oral formulations - fosfomycin. Fosfomycin has a wide spectrum of activity against Gram-positive and Gram-negative bacteria causing neonatal sepsis. It is mainly used for resistant urinary tract infections in adults, but has licenced neonatal and paediatric doses in Europe (though dosing regimens vary between countries). Both oral and IV formulations are available. A large clinical trial to assess the efficacy of a fosfomycin plus an aminoglycoside combination (compared to the current WHO recommended ampicillin and gentamicin) is anticipated, including sites in Kenya. The ultimate aim is for fosfomycin to be included in the WHO Essential Medicines List for children (EMLc) and be available for use in developing countries, where rates of resistance to ampicillin and gentamicin have been estimated at over 40%. The first steps before this trial are to clarify the pharmacokinetics (PK) and safety profile of fosfomycin in neonates, as well as generating further information regarding local patterns of bacterial susceptibility to fosfomycin. The aim of this study is to fulfil both these steps. Fosfomycin (IV and oral) PK will be investigated among 60 babies admitted to hospital and being treated for presumed sepsis; administered alongside the standard antibiotics. Another 60 babies receiving standard treatment only (without PK sampling) will be monitored in the same way to compare adverse events. In the laboratory at CGMR-C, previously archived bacterial isolates will be tested for their sensitivity to fosfomycin.

ELIGIBILITY:
Inclusion Criteria:

* Age 0 to 28 days inclusive
* Weight >1500g
* Born (an estimated) >34 weeks gestation (calculated as per the Ballard Maturational Assessment)
* Admitted to hospital and eligible to receive IV antibiotics, according to national guidelines

Exclusion Criteria:

* Baseline sodium level >= 150mmol/L
* Baseline creatinine >= 150 micromol/L
* Presenting with severe (grade 3) Hypoxic Ischaemic Encephalopathy (HIE), defined as per Sarnat and Sarnat as a stuporous, flaccid infant (with or without seizure activity) with suppressed brainstem and autonomic functions and absent reflexes
* Requiring cardiopulmonary resuscitation on admission
* Jaundice requiring exchange transfusion
* Admitted as a transfer after an overnight inpatient stay at another hospital
* Known allergy or contraindication to fosfomycin
* A specific clinical indication for another class of antibiotic (other than the nationally recommended standard-of-care)
* More than 4 hours after initiating ampicillin plus gentamicin (one dose), which allows for administration of these first-line antibiotics not to be delayed by study procedures
* Concurrent participation in another clinical trial
* Attending clinician's judgement that the child is so severely ill that adequate communication about the study with the parent or legal guardian is not possible.
* Not planning to remain resident in the County for the next 28 days.
* Lack of consent

Max Age: 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Actual)
Dates: Start 2018-03-15 (Actual); Primary Completion 2019-03-14 (Actual); Study Completion 2019-05-24 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic disposition and absorption parameters of IV and oral fosfomycin in neonates with clinical sepsis | Participants will be followed for the duration of enrolment, an expected average of 7 days
  Fosfomycin Clearance (CL)
Pharmacokinetic disposition and absorption parameters of IV and oral | Participants will be followed for the duration of enrolment, an expected average of 7 days
  Fosfomycin Volume of Distribution
Pharmacokinetic disposition and absorption parameters of IV and oral | Participants will be followed for the duration of enrolment, an expected average of 7 days
  Fosfomycin Oral Bioavailability (F)

SECONDARY OUTCOMES:
Difference between the groups in mean 48-hour plasma sodium concentrations | 48 hours
  Biochemistry will be checked at 48 hours for participants in both groups
Difference between the groups in mean 7-day plasma sodium concentrations | 7 days
  Biochemistry will be checked at 7 days for participants in both groups
Difference between groups in the rate of adverse events (any grade) to 28 days after enrolment in the study | from patient randomization to visit D28
  Neonates will be reviewed every day by study clinicians, working together with the hospital team. All adverse events will be documented and reported in both arms.

CONTACTS AND LOCATIONS:
Overall Officials: James A Berkley, Prof, Principal Investigator — KEMRI/Wellcome Trust Research Programme and University of Oxford - UK
Locations (1):
- KEMRI / Wellcome Trust Research Programme, Kilifi, Kenya

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Gastine S, Obiero C, Kane Z, Williams P, Readman J, Murunga S, Thitiri J, Ellis S, Correia E, Nyaoke B, Kipper K, van den Anker J, Sharland M, Berkley JA, Standing JF. Simultaneous pharmacokinetic/pharmacodynamic (PKPD) assessment of ampicillin and gentamicin in the treatment of neonatal sepsis. J Antimicrob Chemother. 2022 Feb 2;77(2):448-456. doi: 10.1093/jac/dkab413. PMID 35107141
- [Derived] Obiero CW, Williams P, Murunga S, Thitiri J, Omollo R, Walker AS, Egondi T, Nyaoke B, Correia E, Kane Z, Gastine S, Kipper K, Standing JF, Ellis S, Sharland M, Berkley JA; NeoFosfo Study Group. Randomised controlled trial of fosfomycin in neonatal sepsis: pharmacokinetics and safety in relation to sodium overload. Arch Dis Child. 2022 Sep;107(9):802-810. doi: 10.1136/archdischild-2021-322483. Epub 2022 Jan 25. PMID 35078765
- [Derived] Kane Z, Gastine S, Obiero C, Williams P, Murunga S, Thitiri J, Ellis S, Correia E, Nyaoke B, Kipper K, van den Anker J, Sharland M, Berkley JA, Standing JF. IV and oral fosfomycin pharmacokinetics in neonates with suspected clinical sepsis. J Antimicrob Chemother. 2021 Jun 18;76(7):1855-1864. doi: 10.1093/jac/dkab083. PMID 33855449